CLINICAL TRIAL: NCT01681134
Title: A Comparison of Effects of Short-Term Steady State Low Dose Exposure of Extended Release (Advagraf®) and Immediate Release (Prograf®) Formulations of Tacrolimus on Renal Perfusion and Function in Healthy Male Volunteers
Brief Title: A Comparison of the Effects of Extended Release Tacrolimus (Advagraf®) vs. Immediate Release Tacrolimus (Prograf®) on Kidney Function in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FKC-016
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: tacrolimus; Advagraf®; Prograf®; Glomerular Filtration Rate; Effective Renal Plasma Flow; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf followed by Prograf (Experimental)
  Interventions: Drug: Advagraf®; Drug: Prograf®
- Prograf followed by Advagraf (Experimental)
  Interventions: Drug: Advagraf®; Drug: Prograf®

INTERVENTIONS:
Drug: Advagraf® — oral
  Other Names: tacrolimus XL, FK506E
Drug: Prograf® — oral
  Other Names: tacrolimus, FK506

SUMMARY:
The purpose of the study is to evaluate the drug profiles (pharmacokinetics) and effects (pharmacodynamics) of Advagraf® and Prograf® on the kidneys.

DETAILED DESCRIPTION:
This is a 2 Period study. In Period 1, subjects will be assigned randomly to receive Advagraf® or Prograf® administered once or twice daily, respectively, for a period of 10 days. In Period 2, subjects will be converted from Advagraf® to Prograf® or from Prograf® to Advagraf® for 10 additional days of dosing. Dose adjustments will be made based on the monitoring of drug levels in blood.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* No previous/current history of infection, cerebrovascular, neurological, cardiovascular, endocrine, pulmonary, immunologic or metabolic disease or significant systemic disease, glucose intolerance, gout or hematological disorder
* Normal 12-lead Electrocardiogram (ECG)
* Systolic blood pressure <140 mm Hg and diastolic blood pressure <90 mm Hg
* Non-smoker within 3 months prior to screening
* Willing to abstain from alcohol during the study

Exclusion Criteria:

* Positive screen for illicit drug or alcohol consumption
* Subject has hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or history of cancer (excluding completely excised squamous or basal cell carcinoma)
* Positive tuberculin skin test or known history of tuberculosis infection
* Known history of serious head injuries, seizures or eating disorders
* Body Mass Index <18.0 or >30.0
* History of renal dysfunction, clinically significant creatinine or clinically significant abnormal liver function tests, hemoglobin <130 g/L
* Plasma donation ≥ 500 mL within 7 days prior to first dose of study drug, donation or whole blood loss 50-499 mL within 30 days or ≥ 499 mL within 56 days prior to first dose of study drug.
* Drug or alcohol abuse within 1 year prior to study entry
* Steroid injections within 12 weeks prior to first dose of study drug
* Live vaccine within 7 days prior to first dose of study drug

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Effective Renal Plasma Flow (ERPF) | up to Day 20
  Estimated by aminohippurate sodium (PAH) clearance

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | Pre-dose (Day -4), Day 10, Day 20
  Estimated by sinistrin clearance

CONTACTS AND LOCATIONS:
Overall Officials: Associate Director, Medical Affairs, Study Director — Astellas Pharma Canada, Inc.
Locations (1):
- INC Research, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Zaltzman JS, Lai V, Schulz MZ, Moon KH, Cherney DZ. A randomized cross-over comparison of short-term exposure of once-daily extended release tacrolimus and twice-daily tacrolimus on renal function in healthy volunteers. Transpl Int. 2014 Dec;27(12):1294-302. doi: 10.1111/tri.12435. Epub 2014 Sep 29. PMID 25160518